CLINICAL TRIAL: NCT05076760
Title: Phase I Study Evaluating MEM-288 Oncolytic Virus Alone and in Combination With Standard of Care Therapy in Advanced Solid Tumors
Brief Title: MEM-288 Oncolytic Virus Alone and in Combination With Standard of Care Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memgen, Inc. (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); Duke Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-2003
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor; Advanced Cancer; Metastatic Cancer; Non Small Cell Lung Cancer; Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma; Melanoma; Pancreatic Cancer; Triple Negative Breast Cancer; Head and Neck Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Carcinoma, Merkel Cell; Melanoma; Pancreatic Neoplasms; Triple Negative Breast Neoplasms; Head and Neck Neoplasms | interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MEM-288 Intratumoral Injection (Complete) (Experimental): Part 1A MEM-288 monotherapy: Patients with accessible, subcutaneous, or superficial lymph node lesion ≥ 1 cm3 that is palpable will receive intratumoral injection of MEM-288 once every 3 week (planned 2 doses, maximum 6 doses) at one of three dose cohort levels.
  * Dose cohort level 1 (1 x 10^10 viral particles)
  * Dose cohort level 2 (3.3 x 10^10 viral particles)
  * Dose cohort level 3 (1 x 10^11 viral particles)
  Interventions: Biological: MEM-288 Intratumoral Injection
- MEM-288 Intratumoral Injection plus anti-PD1 (Nivolumab) Intravenous Infusion (Complete) (Experimental): Part 1B MEM-288 plus nivolumab combination: Patients with accessible, subcutaneous, or superficial lymph node lesion ≥ 1 cm3 that is palpable will receive intratumoral injection of MEM-288 maximum total dose of 1x10^11 viral particles once every 3 week (planned 2 doses, maximum 6 doses). MEM-288 may be injected in multiple lesions until the maximum injection dose (1x10^11 viral particles) is reached (minimum dose per lesion of 1x10^10 viral particles). Nivolumab 360 mg IV every 3 weeks.
  Interventions: Biological: MEM-288 Intratumoral Injection; Biological: Nivolumab
- MEM-288 Intratumoral Injection plus Docetaxel Intravenous Infusion (Open) (Experimental): Part 1C MEM-288 plus docetaxel combination: Patients with advanced NSCLC will be randomized 1:1 to receive either an initial priming dose of MEM-288 (1x10^11 viral particles) injected into an accessible lesion(s) alone (Day 1) followed by MEM-288 in combination with standard of care docetaxel every 3 weeks, with up to 6 doses MEM-288, or MEM-288 injected into an accessible lesion(s) in combination with standard of care docetaxel therapy Day 1 and every 3 weeks up to 6 doses of MEM-288.
  Interventions: Biological: MEM-288 Intratumoral Injection; Drug: Docetaxel

INTERVENTIONS:
Biological: MEM-288 Intratumoral Injection — Intratumoral injection of MEM-288, conditionally replicative oncolytic adenovirus vector encoding transgenes for human interferon beta (IFNβ) and a recombinant chimeric form of CD40-ligand (MEM40).
Biological: Nivolumab — anti-PD1 monoclonal antibody
  Other Names: Opdivo
  Arms: MEM-288 Intratumoral Injection plus anti-PD1 (Nivolumab) Intravenous Infusion (Complete)
Drug: Docetaxel — 75 mg/m2 intravenous administration every 3 weeks
  Arms: MEM-288 Intratumoral Injection plus Docetaxel Intravenous Infusion (Open)

SUMMARY:
This is a multipart, open-label, multi-center dose escalation, dose expansion phase I clinical trial designed to evaluate the safety, tolerability, maximum tolerated dose (MTD), recommended phase 2 dose (RP2D), and preliminary efficacy of MEM-288 in patients with advanced solid tumors. Eligible subjects must have a tumor lesion(s) which is accessible for injection.

The dose escalation phase (Part 1A - advanced solid tumors) has completed and is closed to enrollment. This phase evaluated multiple doses of MEM-288 dosed via intratumoral injection once every 3 weeks to assess safety, tolerability, preliminary efficacy, and to determine the MTD.

The dose expansion phase has multiple parts for advanced NSCLC. Part 1B has completed after evaluation of MEM-288 dosed via intratumoral injection in combination with standard of care nivolumab dosed via intravenous injection.

In a separate dose expansion arm (Part 1C) that is open for enrollment, patients with advanced NSCLC will be randomized to receive either an initial priming dose of MEM-288 injected into an accessible lesion (s) alone (Day 1) followed by MEM-288 in combination with standard of care docetaxel every 3 weeks up to 6 doses or MEM-288 injected into an accessible lesion(s) in combination with standard of care docetaxel therapy Day 1 and every 3 weeks up to 6 doses.

The study rationale is that the oncolytic effect of MEM-288 combined with the presence of CD40L and type 1 IFN in injected tumors will provide a strong signal for DC-mediated T cell activation leading to generation of systemic anti-tumor T cell responses with broad specificity akin to what is observed in the abscopal effect.

DETAILED DESCRIPTION:
MEM-288 is a conditionally replicative oncolytic adenovirus vector encoding transgenes for human interferon beta (IFNβ) and a recombinant chimeric form of CD40-ligand (MEM40). MEM-288 was developed as an immunotherapy for cancer and was engineered to selectively replicate in cancer cells leading to cancer cell lysis but not cytotoxicity towards normal cells. Simultaneously, MEM-288 is designed to stimulate an anti-tumor immune response through expression of its encoded immune agonist transgenes. MEM-288 is designed to provide both antitumor activity as a standalone monotherapy and in combination with other agents to enhance the efficacy of immune checkpoint inhibition or chemotherapy.

This phase I trial is conducted in multiple parts. The first part is an open-label, dose escalation trial of MEM-288 monotherapy in which investigators aim to find the MTD and recommended phase II dose for the planned combination of MEM-288 with an immune checkpoint inhibitor. Patients (≥ 18 years old) eligible for study enrollment include those with either advanced/metastatic NSCLC, cutaneous squamous-cell carcinoma (cSCC), Merkel cell, melanoma, triple negative breast cancer (TNBC), pancreatic cancer, or head and neck cancer, who progressed following previous anti-PD-1/PD-L1 therapy, with a tumor lesion which is accessible for injection. Part 1A has completed and is closed to enrollment.

The primary study objective of the monotherapy dose escalation portion of the study is to determine the safety, tolerability, and maximum tolerated dose (MTD) of intratumoral administration of MEM-288 as a single agent. Secondary objectives will assess efficacy overall response rate, as well as disease control rate, progression free survival, duration of response, and anti-tumor immune responses.

Following completion of Part 1A, there are multiple dose expansion arms designed to test MEM-288 with concurrent therapies for patients with first relapsed or refractory advanced/metastatic NSCLC following front-line anti-PD-1/PD-L1 with or without concurrent chemotherapy.

The primary study objective of the combination portion of the study is to determine the the safety and tolerability of MEM-288 in combination with either nivolumab (Part 1B) or docetaxel (Part 1C).

MEM-288 will be administered via intratumoral injection once every 3 weeks (planned 2 doses, maximum 6 doses) at an assigned dose cohort level (from 1x10^10 to 1x10^11 viral particles) for the Part 1A .

For study Parts 1B and 1C, MEM-288 will be administered via intratumoral injection once every 3 weeks (planned 2 doses, maximum 6 doses) at an assigned dose total dose of 1x10^11 viral particles. MEM-288 may be injected in multiple lesions until the maximum injection dose (1x10^11 viral particles) is reached.

For Part 1B, nivolumab will be administered at a dose of 360 mg via intravenous infusion once every 3 weeks, with optional maintenance nivolumab therapy every 3 weeks for up to 2 years.

For Part 1C, patients with advanced NSCLC will be randomized to receive either an initial priming dose of MEM-288 injected into an accessible lesion (s) alone (Day 1) followed by MEM-288 in combination with standard of care docetaxel every 3 weeks up to 6 doses or MEM-288 injected into an accessible lesion(s) in combination with standard of care docetaxel therapy Day 1 and every 3 weeks up to 6 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and provide informed consent.
2. Willingness and ability to comply with scheduled study visits and procedures.
3. Adult men or women age ≥ 18 years.
4. ECOG performance status of 0 or 1.
5. Part 1A monotherapy: Advanced/metastatic NSCLC, cSCC, Merkel cell, melanoma, TNBC, pancreatic cancer, or head and neck cancer.
6. Parts 1B and 1C combination: Advanced/metastatic NSCLC which has progressed following front-line anti-PD-1/PD-L1 with or without concurrent chemotherapy.
7. Per each tumor type shown below, the specific initial standard of care therapies after which the subjects with specific histologies must have progressed have been included. Subjects will have been treated with at least one or more than one line of therapy prior to enrollment in the study.

   1. Non-small cell lung cancer (NSCLC)

      Part 1A monotherapy
      * Must have progressed on standard therapy, including platinum-based chemotherapy and checkpoint inhibitor therapy (combined or sequential).
      * Patients with tumors that have known actionable molecular alteration such in EGFR, ALK, ROS-1, BRAF, RET, MET, and KRAS must have progressed on standard directed molecular therapy, and platinum-based chemotherapy.

      Part 1B MEM-288 plus nivolumab combination
      * Must have first progression more than (>) 84 days following initiation (cycle 1 day 1) of their most recent anti-PD-1 or PD-L1 checkpoint inhibitor therapy with or without concurrent chemotherapy

      Part 1C MEM-288 plus docetaxel combination must have either:
      * first progression with anti-PD-1 or PD-L1 checkpoint inhibitor therapy with or without concurrent chemotherapy, or
      * progressed following initial first line anti-PD-1 or PD-L1 monotherapy followed by 2nd line platinum chemotherapy (with or without continuation of their first line anti-PD-1 or PD-L1 therapy).
   2. Cutaneous squamous-cell carcinoma (cSCC)

      * Must have progressed on standard therapy, including platinum-based chemotherapy and/or checkpoint inhibitor therapy.
   3. Merkel cell Carcinoma

      * Must have progressed on standard checkpoint inhibitor therapy.
   4. Melanoma

      * Subjects must have received a BRAF inhibitor as monotherapy or in combination with other targeted agents for BRAF V600E mutant melanoma.
      * Subjects must have received an anti-PD-1/ PD-L1inhibitor as monotherapy or combination with anti-CTLA-4 inhibitor or other therapies.
   5. Pancreatic cancer

      * Progression after systemic chemotherapy which included either gemcitabine or Fluorouracil (5-FU)-based regimen (including capecitabine).
   6. Triple negative breast cancer (TNBC)

      * Prior treatment (for advanced, metastatic or (neo)adjuvant) must have included a taxane and/or anthracycline-based therapy.
   7. Head and Neck Cancer

      * Prior treatment requirement in the metastatic or unresectable locally advanced setting include:
      * Subjects must have received a platinum containing chemotherapy regimen for treatment of primary tumor in locally advanced, or metastatic settings
      * Subjects must have received an anti-PD-1/ PD-L1 as monotherapy or in combination with chemotherapy.
8. Progressed following therapy with at least one PD-1 or PD-L1 checkpoint inhibitor (regardless of PD-L1 expression status), except for patients with pancreatic cancer.

   a) Prior progression on a PD-1 or PD-L1 checkpoint inhibitor should be unequivocal; progression that occurs within the first 8 weeks of treatment on these agents should be confirmed with a second CT at least 4 weeks apart (to exclude pseudo-progression).
9. Patients with activating EGFR mutation or ALK rearrangement which is expected to be responsive to available tyrosine kinase inhibitor therapy, must have been previously treated with an applicable tyrosine kinase inhibitor.
10. Tumor lesion which is deemed feasible for biopsy and injection under CT or ultrasound guidance (based on size, location, and visibility) by an interventional radiologist, and patient willing and able to provide tissue from biopsy of this lesion. Injected tumor should be > 1 cm3 in volume and should not encase or be inseparable from vital structures such as major nerves or blood vessels.

    a) For Part 1 monotherapy patients treated at the first dose level, the tumor for injection must be an accessible cutaneous, subcutaneous, or superficial lymph node lesion that is palpable.
11. Measurable disease, as defined per RECIST version 1.1.
12. Prior history of brain metastases are eligible, provided:

    1. Brain metastases have been treated
    2. Asymptomatic from the brain metastases
    3. Corticosteroids prescribed for the management of brain metastases have been discontinued at least 7 days before registration to study
    4. Brain metastases are stable on pre-registration imaging
    5. No evidence of leptomeningeal disease
13. Life expectancy > 3 months.
14. Adequate organ and marrow function as defined below:

    1. Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
    2. Hemoglobin ≥90 g/L (or ≥9 g/dL)
    3. Platelets ≥100 x 10^9/L
    4. Calculated creatinine clearance of >50 mL/min using Cockcroft Gault equation
    5. Total bilirubin ≤ 1.5 x institutional upper limit of normal
    6. AST (SGOT) and ALT (SGPT) ≤2.5 x institutional upper limit of normal
    7. If Alkaline Phosphatase ≥ 2.5 x institutional upper limit of normal, then AST and ALT must be ≤ 1.5 x institutional upper limit of normal
15. Patients of childbearing age must not be pregnant and must use established contraceptive strategies:

    1. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
    2. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
    3. Male subjects should agree to use an adequate method of barrier contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Pregnant or breast feeding.
2. Serious uncontrolled medical disorder, psychiatric condition or laboratory abnormalities that, in the opinion of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
3. Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic), or significant traumatic injury, within 4 weeks prior to starting study treatment or has not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy are exceptions and patients can receive study treatment ≥1 week after these procedures.
4. History of clinically significant noninfectious interstitial pneumonitis (i.e., limiting activities of daily living or requiring therapeutic intervention), including clinically significant radiation pneumonitis.
5. Residual toxicity from prior anticancer therapy of grade 3 or greater (CTCAE v5.0), with the exception of alopecia.
6. Concurrent use of other anticancer approved or investigational agents.
7. Clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

   1. unstable angina within 6 months prior to screening
   2. myocardial infarction within 6 months prior to screening
   3. history of documented congestive heart failure (New York Heart Association functional classification III-IV)
   4. cardiac arrhythmias not controlled with medication
8. Active autoimmune disease requiring disease modifying therapy (except vitiligo, Grave's, or psoriasis not requiring systemic treatment).
9. Any form of active primary or secondary immunodeficiency.
10. Receiving ≥10 mg daily prednisone (or equivalent).
11. Prior malignancy (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, cervical/dysplasia endometrial, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required or anticipated to be required during the study period.
12. Active systemic infections requiring intravenous antibiotics.
13. Prior therapy with anti-tumor vaccines or other immune-stimulatory antitumor agents (other than FDA approved and National Comprehensive Cancer Network [NCCN] recommended systemic therapies).
14. Prisoners or subjects who are involuntarily incarcerated, or who are compulsorily detained for treatment of either a psychiatric or physical illness.
15. Any unresolved grade 2 irAE (except adequately treated endocrine irAE).
16. Any toxicity that led to permanent discontinuation of prior anti-PD-1/PD-L1 immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Part 1A Monotherapy: Maximum Tolerated Dose (MTD) | 21 days
  MTD is defined as the highest dose with ≤ 17% dose limiting toxicity (DLT) rate.
Safety and Tolerability assessed by Adverse Events (AEs) | 4.5 months
  An adverse event (AE) is any untoward medical occurrence in a subject receiving study drug and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended or worsening sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to use of the study drug.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 39 weeks
  ORR measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Disease Control Rate (DCR) | up to 39 weeks
  DCR measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Progression Free Survival (PFS) | up to 5 years
  To determine the PFS days post treatment initiation.
Overall Survival (OS) | up to 5 years
  To determine the survival days post treatment initiation.

OTHER OUTCOMES:
Exploratory Biomarker Analysis | 4.5 months
  Analysis of potential associations between biomarker measures and anti-tumor activity, immunogenicity, and immune-activation assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, MD, PhD, Principal Investigator — Duke Cancer Institute; Andreas Saltos, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Duke Cancer Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Memgen, Inc. is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission.
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.